CLINICAL TRIAL: NCT01334814
Title: Chronic Versus Intermittent Deep Brain Stimulation for Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Ryan J. Uitti, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1324-02
Record Dates: First submitted 2010-03-09; First posted 2011-04-13 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Deep Brain Stimulation (Model 7438 Therapy Controller) — Deep brain stimulation (DBS) is a surgical procedure used to treat a variety of disabling neurological symptoms
  Other Names: Model 7438 Therapy Controller

SUMMARY:
The proposed study is a randomized, single blind trial of intermittent versus continuous stimulation among essential tremor (ET) patients with a chronic history of continuous stimulation.

DETAILED DESCRIPTION:
The proposed study is a randomized, single blind trial of intermittent versus continuous stimulation among essential tremor (ET) patients with a chronic history of continuous stimulation. The trial is 10 weeks in length with clinical evaluations (about 60 minutes) performed on weeks 1, 2, 6, and 10, and phone interviews (about 5 minutes) on weeks 3, 4, 5, 7, 8, and 9. The study includes outcome measures of tremor, stimulation-induced side effects, sleep quality, and voltage threshold for optimal tremor control and sustained side-effects.

ELIGIBILITY:
Inclusion Criteria:

* individuals with essential tremor who are at least 6 months status-post thalamic stimulator placement
* maintained a consistent chronic or intermittent stimulation schedule for at least 4 consecutive weeks prior to study enrollment
* no changes in stimulation parameters for at least 2 consecutive months prior to study enrollment

Exclusion Criteria:

* patients with clinically significant dementia (i.e., a score less than 24 out of 30 on the Mini Mental Status Exam14)
* women who are not post-menopausal
* patients with other significant neurological or psychiatric disease other than essential tremor
* patients treated with pallidotomy or thalamotomy
* patients with significant psychiatric disturbance as determined by Diagnostic and Statistical Manual-IV criteria which would make informed consent/cooperation problematic

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2002-01; Primary Completion 2005-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
sleep quality | 10 weeks
  The trial is 10 weeks in length with clinical evaluations (about 60 minutes) performed on weeks 1, 2, 6, and 10, and phone interviews (about 5 minutes) on weeks 3, 4, 5, 7, 8, and 9.

SECONDARY OUTCOMES:
measures of tremor,voltage threshold for optimal tremor control | 10 weeks
Side effects | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Uitti, MD, Principal Investigator — Mayo Clinic